CLINICAL TRIAL: NCT01858896
Title: Hypoglycemia Associated Autonomic Dysfunction
Brief Title: GLP-1 and Hypoglycemia
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Chairman of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP00055308
Record Dates: First submitted 2013-05-13; First posted 2013-05-21 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: hypoglycemia; GLP-1; Type 2 diabetes; endothelial function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucagon-Like Peptide -1 (GLP-1) infusion (Active Comparator): Infusion of GLP-1 during experimental period
  Interventions: Drug: Glucagon-Like Peptide- 1 (GLP-1) infusion
- Saline Infusion (Placebo Comparator): Saline infusion during experimental period
  Interventions: Other: Placebo Comparator: Saline Infusion

INTERVENTIONS:
Drug: Glucagon-Like Peptide- 1 (GLP-1) infusion — GLP-1 infusion during experimental period
  Other Names: GLP-1
  Arms: Glucagon-Like Peptide -1 (GLP-1) infusion
Other: Placebo Comparator: Saline Infusion — Saline infusion (placebo) during experimental period
  Other Names: Saline infusion
  Arms: Saline Infusion

SUMMARY:
Low blood sugar can negatively affect how blood vessels function, and this can lead to an increase in the risk for heart attacks, strokes and other problems related to the stiffening and blockage of blood vessels. The purpose of this study is to learn if and how glucagon-like peptide-1 (GLP-1; a naturally occurring hormone in the gut) changes the effects that low blood sugar levels have on blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* 14 (7 males, 7 females) healthy controls age 30-60 yr.
* 14 (7 males, 7 females) people with type 2 DM age 30-60 yr.
* For type 2 DM: HbA1c 6-10.0%
* No significant diabetic tissue complications (i.e. history of retinopathy, neuropathy, stasis ulcers, etc.)
* Body mass index >25kg • m-2

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Plasminogen Activation inhibitor-1 (PAi-1) | change from baseline to end of clamp period
  measurements of change in PAi-1 at baseline and during the end of the glucose clamp period (2 hours)
Change in Flow mediated dilation (FMD) | change from baseline and end of clamp
  flow mediated dilation of the brachial artery will be measured for change from baseline and end of glucose clamp (~4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N Davis, MBBS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States